CLINICAL TRIAL: NCT02893631
Title: Assessment of Hemostasis Disorders in Tissue Plasminogen Activator Treated (rtPA-treated) Patients Requiring Endovascular Treatment for Ischemic Stroke
Brief Title: Assessment of Hemostasis Disorders in rtPA-treated Patients Requiring Endovascular Treatment for Ischemic Stroke
Acronym: HEMOLYSE
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: AGR_2015_25
Record Dates: First submitted 2016-08-31; First posted 2016-09-08 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
Stroke treatment includes thrombolysis, thrombectomy for patients with proximal artery occlusion and sometimes neurosurgery. It rises questions regarding hemostasis: thrombolysis induces fibrinolysis but its effects on coagulation, fibrinogen and platelets and duration of these effects are unknown. Thus management of antithrombotics and hemostasis during thrombectomy and surgery is an issue.

Objectives : to describe thrombolysis-induced hemostatic disorders (fibrinolysis, coagulation, fibrinogen, platelets) in patients requiring thrombectomy for stroke and to evaluate the time required for the normalization of these disorders.

Methods : Observational monocentric study including rtPA-treated patients requiring endovascular treatment for stroke. Blood sampling within the first 48 hours after rtPA administration to assess of fibrinolysis, coagulation and platelet functions with point of care devices and specific laboratory tests. Record of clinical and biological data.

ELIGIBILITY:
Inclusion Criteria:

* patient over 18
* treatment with rtPA for an acute stroke
* endovascular treatment required

Exclusion Criteria:

* opposition to participate in the study
* long term anticoagulant-treated patient
* pregnant patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: rtPA-treated patients requiring endovascular treatment for ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
fibrinolysis activity | until normalization of fibrinolytic activity, up to 48 hours
  Time required for normalization of fibrinolysis

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claire NGHE, MD, PhD, Principal Investigator — Fondation OPH A de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, France